CLINICAL TRIAL: NCT04546152
Title: Prospective Observational Clinical Trial for Safety and Efficacy of HYAPROF® SOFT and HYAPROF® BALANCE
Brief Title: Safety and Efficacy of the HA-based Dermal Fillers HYAPROF® SOFT and HYAPROF® BALANCE
Acronym: PMCF_HYAPROF
Status: Completed | Type: Observational
Sponsor: BioSCIENCE GmbH (Industry)
Collaborators: HeiMed (Unknown)
Responsible Party: Sponsor
Other Study IDs: CIP HYAPROF SOFT and BALANCE
Record Dates: First submitted 2020-08-26; First posted 2020-09-11 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Dermal Filler
Keywords: Volume Replacement; Facial Filler; Soft Tissue Filler; Hyaluronic Acid

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- HYAPROF® SOFT: HYAPROF® SOFT is indicated for volume replacement (filling of folds), fine to medium folds, lip augmentation, periorbital region.
  Interventions: Device: HYAPROF® SOFT and HYAPROF® BALANCE
- HYAPROF® BALANCE: HYAPROF® BALANCE is indicated for volume replacement (filling of folds), deep folds, nasolabial folds, cheek area, glabella folds. It is not intended for injection to the periorbital region (eyelid, crow's feet, circles under the eyes).
  Interventions: Device: HYAPROF® SOFT and HYAPROF® BALANCE

INTERVENTIONS:
Device: HYAPROF® SOFT and HYAPROF® BALANCE — Dermal filler injection to different facial areas

SUMMARY:
Purpose of this study is the demonstration of safety and efficacy of the dermal fillers HYAPROF® SOFT and HYAPROF® BALANCE for restoration of the facial volume and contour.

DETAILED DESCRIPTION:
This is a prospective, multicenter, observational, open label, two-arm, crossover, PMCF clinical trial for demonstration of the safety and efficacy of the HA-based dermal fillers HYAPROF® SOFT and HYAPROF® BALANCE for restoration of the facial volume and contour. Besides safety aspects, evaluated immediately after the treatment, 4 weeks, 3 and 6 months after the treatment, the performance of the demal fillers are evaluated in the 3 and 6 months follow-up by using GAIS and WSRS.

ELIGIBILITY:
Inclusion Criteria:

* subjects intended for the treatment with HYAPROF® SOFT and/or BALANCE according to the instructions for use of the product
* decision for the treatment with HYAPROF® SOFT and/or BALANCE was made before the subject was recruited for the clinical trial
* subjects signed written informed consent
* adult subjects at least 18 years old
* all Fitzpatrick skin types
* area treated either with HYAPROF® SOFT or HYAPROF® BALANCE - no combination of the products in one treated area

Exclusion Criteria:

* tendency to hypertrophic and keloid scarring
* intolerance to gram-positive bacteria
* prone to active inflammatory or infectious processes
* suffering from acute or chronic skin diseases
* undergoing anti-coagulant therapy
* known allergy to hyaluronic acid
* suffering from autoimmune diseases
* multiple allergies
* pregnancy or lactating women
* subjects unlikely to cooperate in the clinical investigation or to comply with the treatment or with the clinical investigation visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects intended for the treatment with HYAPROF® SOFT and BALANCE according to the instructions for use of the products.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2022-01-22 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Global aesthetic improvement 3 months | 3 months
  Global aesthetic improvement assessment acc. to the Global Aesthetic Improvement Scale (GAIS); 3: very much improved, 2: much improved, 1: improved, 0 unchanged, -1: worse
Global aesthetic improvement 6 months | 6 months
  Global aesthetic improvement assessment acc. to the Global Aesthetic Improvement Scale (GAIS); 3: very much improved, 2: much improved, 1: improved, 0 unchanged, -1: worse
Wrinkle severity assessment 3 months | 3 months
  Wrinkle severity assessment acc. to the Wrinkle Severity Rating Scale (WSRS); 1: wrinkles absent, 2: slight wrinkles, 3: moderate wrinkles, 4: severe wrinkles, 5: very severe wrinkles
Wrinkle severity assessment 6 months | 6 months
  Wrinkle severity assessment acc. to the Wrinkle Severity Rating Scale (WSRS); 1: wrinkles absent, 2: slight wrinkles, 3: moderate wrinkles, 4: severe wrinkles, 5: very severe wrinkles
Number of subjects with wrinkle severity improvement 3 months | 3 months
  Number of subjects with at least one scale point improvement in the wrinkle severity assessment (WSRS) with respect to baseline
Number of subjects with wrinkle severity improvement 6 months | 6 months
  Number of subjects with at least one scale point improvement in the wrinkle severity assessment (WSRS) with respect to baseline

SECONDARY OUTCOMES:
Product safety immediately after the treatment | Immediately after the treatment
  Side effects and adverse event recording; degree of severity: mild, moderate, severe
Product safety 4 weeks | 4 weeks
  Side effects and adverse event recording; degree of severity: mild, moderate, severe; duration of the event
Product safety 3 months | 3 months
  Side effects and adverse event recording; degree of severity: mild, moderate, severe; duration of the event
Product safety 6 months | 6 months
  Side effects and adverse event recording; degree of severity: mild, moderate, severe; duration of the event

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - BioSCIENCE Investigation Site #01, Bad Honnef
  - BioSCIENCE Investigation Site #02, Kempten

IPD SHARING:
Plan to Share IPD: No